CLINICAL TRIAL: NCT03435783
Title: Brief Electronic Intervention for Heavy Drinking and Sex Risk Among MSM Seeking HIV Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Tyler Wray, Assistant Professor, Brown University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 1411001155
Record Dates: First submitted 2017-08-02; First posted 2018-02-19 (Actual); Results first posted 2019-04-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: HIV Infections; Alcohol Abuse
MeSH Terms: conditions — HIV Infections; Alcoholism

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial where participants are assigned to either a treatment or control group.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Brief Electronic Intervention
- Attention-matched control (Active Comparator)
  Interventions: Behavioral: Attention-Matched Control

INTERVENTIONS:
Behavioral: Brief Electronic Intervention — The brief electronic intervention will allow users to receive normative feedback based on their alcohol use and sexual activity. Users who show interest in changing their behavior will also be asked to create a plan to do so.
  Arms: Intervention
Behavioral: Attention-Matched Control — Participants will view a video clip on general health promotion that is a similar length as the intervention arm.
  Arms: Attention-matched control

SUMMARY:
The overall objective of this research is to use both qualitative and quantitative data to inform the development of a technology-based intervention for heavy drinking and sexual risk behavior among men who have sex with men (MSM) who are seeking free HIV testing. Investigators will be conducting a randomized-controlled pilot test of the intervention among MSM seeking HIV testing in community-based settings to explore its potential impact on alcohol and HIV-related behavioral outcomes. This research will ultimately produce a combined, theory-based, and technology- delivered intervention for heavy drinking and sex risk that is fully portable and has been preliminarily tested for efficacy in community settings where high-risk MSM engage with prevention services.

ELIGIBILITY:
Inclusion Criteria:

1. Biologically male
2. Aged 18 or older
3. Fluent English speaker
4. Unprotected anal sex with a casual male partner at least once in the past 3 months
5. Heavy alcohol use during the past 2-weeks (>14 drinks per week, or at least one occasion of 5+ drinks on a given occasion)
6. Breath alcohol concentration (BrAC) of .000 at the time of enrollment
7. No history of complex alcohol withdrawal
8. HIV-negative

Exclusion Criteria:

1. Individuals who are HIV-positive
2. Individuals who participated in other phases of the research
3. Individuals who report being coerced to participate

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2018-03-03 (Actual); Study Completion 2018-03-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brown University School of Public Health, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Post-test Counseling (Control): Participants will receive standard post-test counseling alone. This counseling consists of a one-on-one session with a Bachelor's level counselor and involves identifying personal risks for HIV, discussing options for reducing that risk, and eliciting commitment to a plan in order to reduce future risk.
- Brief Web-based Intervention: This web-based intervention will be delivered on a tablet, and will involve presenting feedback on HIV risk behavior and alcohol use, normative comparisons with other gay/bi men in their age group, exercises designed to help them reflect on whether or not they want to make a change, and change planning modules to help users select an option that works for them and get them started.
Period: Overall Study
Arm/Group | Standard Post-test Counseling (Control) | Brief Web-based Intervention
Started | 20 | 20
Completed | 20 | 19
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Attention-matched Control | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.7 (8.3) | 28.8 (9.9) | 28.3 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 20 | 20 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 17 | 19 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 15 | 13 | 28
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of New Sex Partners, Past 30 Days
Description: Assessed via self-report using Timeline Follow Back (TLFB)
Time Frame: Past 30 days
Measure: Mean (Standard Deviation); unit: New partners
Arm/Group | Standard Post-test Counseling (Control) | Brief Web-based Intervention
Number analyzed (Participants) | 20 | 20
New partners | 2.53 (3.6) | 1.37 (1.2)

2. Primary Outcome: Number of Condomless Anal Sex Events, Past 30 Days
Description: Assessed via self-report using Timeline Follow Back (TLFB); count of the number of such events.
Time Frame: Past 30 days
Measure: Mean (Standard Deviation); unit: Events
Arm/Group | Standard Post-test Counseling (Control) | Brief Web-based Intervention
Number analyzed (Participants) | 20 | 20
Events | 1.06 (1.6) | 1.08 (1.3)

3. Primary Outcome: Number of Drinking Days, Past 30 Days
Description: Assessed via self-report using Timeline Follow Back (TLFB); count of the average number of drinking days in the past 30
Time Frame: Past 30 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Standard Post-test Counseling (Control) | Brief Web-based Intervention
Number analyzed (Participants) | 20 | 20
Days | 10.8 (6.9) | 7.04 (5.0)

4. Primary Outcome: Number of Heavy Drinking Days (5 or More), Past 30 Days
Description: Assessed via self-report using Timeline Follow Back (TLFB); count of the number of days.
Time Frame: Past 30 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Standard Post-test Counseling (Control) | Brief Web-based Intervention
Number analyzed (Participants) | 20 | 20
Days | 3.83 (3.6) | 2.67 (1.8)

5. Primary Outcome: Average Number of Drinks Per Drinking Day
Description: Assessed using Timeline Follow Back (TLFB)
Time Frame: Past 30 days
Measure: Mean (Standard Deviation); unit: Drinks
Arm/Group | Standard Post-test Counseling (Control) | Brief Web-based Intervention
Number analyzed (Participants) | 20 | 20
Drinks | 4.73 (2.3) | 4.54 (1.6)

ADVERSE EVENTS:
Time Frame: 3 months (the duration of the study period for all participants).
Arm/Group | Standard Post-test Counseling (Control) | Brief Web-based Intervention
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-07-21): https://cdn.clinicaltrials.gov/large-docs/83/NCT03435783/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-21): https://cdn.clinicaltrials.gov/large-docs/83/NCT03435783/SAP_001.pdf